CLINICAL TRIAL: NCT06661005
Title: Nitrous Oxide for Pain Management During In-Office Gynecology Procedures
Acronym: NO2
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study team didn't have the nitrous oxide to conduct the study.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008947582
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Nitrous Oxide
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: The patient will be consented for the study at their office visit when the decision is made to schedule them for a procedure meeting inclusion criteria for our study. After the patient is consented, they will be randomized to either nitrous oxide or IV sedation. Depending on their randomization group, they will be scheduled on a "Nitrous Day" or an "IV Sedation Day".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrous Day (Experimental): The Nitrous group will receive instructions to arrive at clinic 30 minutes before her procedure in order to sign consent forms. She will not be given instructions to remain NPO and will not be required to have someone bring her to and from the appointment. No IV will be placed. Anesthesia induction will be done by an anesthesiologist with a nitrous oxygen mixture at a 70:30 ratio
  Interventions: Drug: Nitrous oxide
- IV Sedation Day (Active Comparator): The IV sedation group will receive instructions to arrive at clinic 1 hour before her procedure in order to sign consent forms and have an IV placed. She will be given instructions to remain NPO status at least 8 hours prior to the procedure and will need someone to bring her to and from the appointment. Anesthesia induction will be done by an anesthesiologist with propofol per standard protocol.
  Interventions: Drug: IV Sedation

INTERVENTIONS:
Drug: Nitrous oxide — The Nitrous oxide group will receive instructions to arrive at clinic 30 minutes before her procedure in order to sign consent forms. She will not be given instructions to remain NPO and will not be required to have someone bring her to and from the appointment. No IV will be placed. Anesthesia induction will be done by an anesthesiologist with a nitrous oxygen mixture at a 70:30 ratio
  Arms: Nitrous Day
Drug: IV Sedation — Anesthesia induction will be done by an anesthesiologist with propofol per standard protocol. A pulse oximeter will be placed and oxygen will be administered through a nasal cannula and the patient will be instructed to breath.
  Arms: IV Sedation Day

SUMMARY:
The purpose of this study is to evaluate the pain control, patient satisfaction, and efficiency of nitrous oxide used for anesthesia during in-office gynecologic procedures compared to IV sedation. IV sedation for office-based gynecology procedures provides effective anesthesia but requires a recovery time, IV placement, and a ride provided for the patient. Nitrous oxide can be a viable alternative to IV sedation while also reducing recovery time and omitting the need for an IV, NPO status, and a ride home.

DETAILED DESCRIPTION:
Many hysteroscopic procedures require only minimal sedation in order to accomplish adequate pain control and sufficient anesthesia for completion of the procedure. In order to avoid the higher costs and time associated with hospital-based procedures, there is a growing trend to complete these procedures in an office-based setting with IV sedation. With IV sedation, the patients are required to have a ride to and from the appointment, maintain an NPO status for at least 8 hours prior to the appointment, receive proper IV placement prior to the procedure, and remain in the recovery area until anesthesia has worn off, which can take 30 minutes to 1 hour. Several studies in the family planning literature have shown promising results using nitrous oxide for anesthesia during simple in-office procedures such as ****. One pilot study from Madrid demonstrated superior pain control with nitrous oxide when compared to ****.

We believe that nitrous oxide can be a safe, effective, and favorable method for anesthesia for quick and simple office-based gynecologic procedures. Not only will nitrous oxide provide an equal level of pain control, but it also provides several benefits to the patient and the physician. Using nitrous oxide will not require the patient to withstand an uncomfortable IV placement, to maintain NPO status prior to the procedure, or to coordinate a ride before and after the procedure. For the physician, using nitrous oxide for procedures will provide quicker recovery times, allowing physicians to potentially provide services to more patients within a single clinic day.

Nitrous oxide (N2O) was first isolated in 1772 by the English chemist Joseph Priestly and was later discovered to have analgesic properties by Humphry Davy almost twenty years later (Boyle, Goerig, Huang, Priestly). Its role as an analgesic did not take hold until 1863 when Gardner Quincy Colton established the use of nitrous oxide for dental procedures. After its introduction to dentistry, N2O soon became a popular form of pain management in both obstetrics and surgery (Goerig, Huang, Smith).

Nitrous oxide, when inhaled, has both analgesic and anesthetic properties. The exact anesthetic mechanism of action is not completely understood but is thought to be due to non-competitive inhibition of the excitatory NMDA subtype glutamate receptors (Jevtovic). Nitrous oxide provides analgesia by stimulating opioid receptors in the periaqueductal gray matter and noradrenergic receptors in the brainstem, causing a release of endogenous opioids. This release of endogenous opioids dis-inhibits noradrenergic neurons in the brainstem by inhibiting the inhibiting GABA receptors. Consequently, norepinephrine is released into the spinal cord, thereby inhibiting pain signaling (Fujinaga, Sanders).

Although nitrous oxide has been documented as a safe and effective method for pain relief in many areas of medicine, specifically obstetrics, little research exists about its use for pain management for in-office gynecologic procedures. One study by Singh et al evaluated the role of Nitrous Oxide vs no intervention for IUD insertion in nulliparous women and found that nitrous oxide did not reduce pain (Singh). A pilot study by Rubido et al examined nitrous oxide versus no intervention versus paracervical block in women undergoing hysteroscopic polypectomy and found that nitrous oxide outperformed both the control group and paracervical group (Rubido). A third randomized controlled trial studied the superiority of nitrous oxide versus oral analgesia and discovered that nitrous oxide significantly reduced pain scores compared to the control group (Schneider). The purpose of this study is to examine the non-inferiority of nitrous oxide to intravenous sedation for pain management during in-office gynecologic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Negative UPT
* English speaking,
* At the Banner Women's Institute who are consented for any of the following procedures with sedation: Diagnostic hysteroscopy, Hysteroscopic endometrial biopsy, Hysteroscopy, IUD placement, Hysteroscopic IUD removal, Colposcopy, LEEP

Exclusion Criteria:

* Chronic narcotic use,
* Contraindications to Nitrous oxide (i.e. Vit B12 deficiency, pulmonary disease),
* Indication for general anesthesia in the main operating room
* BMI >40
* Non-English Speaking

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — These are female Gynecology patients
Enrollment: 3 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation | Procedure start time to procedure end time.
  Post procedure, patients will be asked to rate their pain using the VASscale, with 0 indicating no pain, to 10 indicating worst possible, unbearable, excruciating pain.
Patient Satisfaction | Procedure start time to procedure end time.
  Post procedure, patients will be asked to rate their satisfaction using the following scale: Very dissatisfied, Dissatisfied, Neutral, Satisfied, or Very Satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyle HE. NITROUS OXIDE: HISTORY AND DEVELOPMENT. Br Med J. 1934 Jan 27;1(3812):153-5. doi: 10.1136/bmj.1.3812.153. No abstract available. PMID 20778037
- [Background] Fujinaga M, Maze M. Neurobiology of nitrous oxide-induced antinociceptive effects. Mol Neurobiol. 2002 Apr;25(2):167-89. doi: 10.1385/MN:25:2:167. PMID 11936558
- [Background] Goerig M, Esch JSA. History of nitrous oxide-with special reference to its early use in Germany. Best Practice & Research Clinical Anaesthesiology. 2001;15(3):313-338.
- [Background] Huang C, Johnson N. Nitrous Oxide, From the Operating Room to the Emergency Department. Curr Emerg Hosp Med Rep. 2016;4:11-18. doi: 10.1007/s40138-016-0092-3. Epub 2016 Mar 22. PMID 27073749
- [Background] Jevtovic-Todorovic V, Todorovic SM, Mennerick S, Powell S, Dikranian K, Benshoff N, Zorumski CF, Olney JW. Nitrous oxide (laughing gas) is an NMDA antagonist, neuroprotectant and neurotoxin. Nat Med. 1998 Apr;4(4):460-3. doi: 10.1038/nm0498-460. PMID 9546794
- [Background] Del Valle Rubido C, Solano Calvo JA, Rodriguez Miguel A, Delgado Espeja JJ, Gonzalez Hinojosa J, Zapico Goni A. Inhalation analgesia with nitrous oxide versus other analgesic techniques in hysteroscopic polypectomy: a pilot study. J Minim Invasive Gynecol. 2015 May-Jun;22(4):595-600. doi: 10.1016/j.jmig.2015.01.005. Epub 2015 Jan 14. PMID 25596171
- [Background] Sanders RD, Weimann J, Maze M. Biologic effects of nitrous oxide: a mechanistic and toxicologic review. Anesthesiology. 2008 Oct;109(4):707-22. doi: 10.1097/ALN.0b013e3181870a17. PMID 18813051
- [Background] Schneider EN, Riley R, Espey E, Mishra SI, Singh RH. Nitrous oxide for pain management during in-office hysteroscopic sterilization: a randomized controlled trial. Contraception. 2017 Mar;95(3):239-244. doi: 10.1016/j.contraception.2016.09.006. Epub 2016 Sep 9. PMID 27621048
- [Background] Singh RH, Thaxton L, Carr S, Leeman L, Schneider E, Espey E. A randomized controlled trial of nitrous oxide for intrauterine device insertion in nulliparous women. Int J Gynaecol Obstet. 2016 Nov;135(2):145-148. doi: 10.1016/j.ijgo.2016.04.014. Epub 2016 Jul 16. PMID 27481016
- [Background] Smith W. Under the influence. A history of nitrous oxide and oxygen Anesthesia. Park Ridge: The Wood Library Museum of Anesthesiology; 1982